CLINICAL TRIAL: NCT06256289
Title: Efficacy of Canagliflozin Versus Metformin in Women With Polycystic Ovary Syndrome Combined With Non-Alcoholic Fatty Liver Disease: A Single-center, Open-labeled Prospective Randomized Controlled
Brief Title: Efficacy of Canagliflozin Versus Metformin in Women With Polycystic Ovary Syndrome
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ping Li,MD (Other)
Responsible Party: Sponsor-Investigator, Ping Li,MD, Principal investigator, The First Affiliated Hospital of Shanxi Medical University
Organization: The First Affiliated Hospital of Shanxi Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FirstofShanxiMU
Record Dates: First submitted 2024-01-28; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Polycystic Ovary Syndrome; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Polycystic Ovary Syndrome; Non-alcoholic Fatty Liver Disease | interventions — Canagliflozin; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- canagliflozin plus metformin group (Experimental): canagliflozin 100 mg once daily plus metformin 1000 mg twice daily
  Interventions: Drug: Canagliflozin 100mg Tab; Drug: Metformin Hydrochloride
- metformin group (Active Comparator): metformin 1000 mg twice daily
  Interventions: Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Canagliflozin 100mg Tab — Canagliflozin 100mg once daily combined Metformin 1000mg twice daily
  Other Names: Invokana
  Arms: canagliflozin plus metformin group
Drug: Metformin Hydrochloride — Metformin 1000mg twice daily
  Other Names: Glucophage

SUMMARY:
The goal of this clinical trial is to investigate the use of ultra-high performance liquid chromatography-mass spectrometry for metabolomics and proteomics research in patients with Polycystic Ovary Syndrome (PCOS) and Non-Alcoholic Fatty Liver Disease (NAFLD). The main questions it aims to answer are:

* How can this technology help identify specific biomarkers for diagnosing PCOS combined with NAFLD?
* What is the role of Canagliflozin in improving the safety and efficacy of treatment for PCOS and NAFLD patients?

Participants, who are 50 non-diabetic women with PCOS, will undergo a series of assessments including cardiovascular metabolic indicators, liver NAFLD screening risk stratification, and insulin resistance index. They will be compared with 50 age and BMI-matched healthy controls. The participants will be randomized to receive either CANA/MET (Canagliflozin 100 mg daily plus Metformin 1000 mg twice daily) or MET (Metformin 1000 mg twice daily) for a continuous period of three months. The study will evaluate various parameters including menstrual patterns, anthropometric parameters, gonadal parameters, glucose-lipid homeostasis, liver enzyme indices, non-invasive hepatic fat changes, metabolomics, and NAFLD-related indicators.

DETAILED DESCRIPTION:
Objective: 1. This study employs the latest ultra-high performance liquid chromatography-mass spectrometry platform for metabolomics and proteomics research to analyze serum samples from patients with Polycystic Ovary Syndrome (PCOS) coexisting with Non-Alcoholic Fatty Liver Disease (NAFLD). The aim is to identify specific biomarkers for the diagnosis of PCOS combined with NAFLD. At the same time, this study explores the pathogenesis and potential new therapeutic targets of PCOS combined with NAFLD at the protein and metabolic levels. 2. The study examines the role of Canagliflozin in improving the safety and efficacy of PCOS and NAFLD patients, providing evidence for the use of SGLT2 inhibitors as an effective treatment for PCOS with NAFLD.

Methods: The study enrolled 50 non-diabetic PCOS women and assessed cardiovascular metabolic indicators including liver NAFLD screening risk stratification, insulin resistance index, etc. These were compared with 50 age and BMI-matched healthy controls. Utilizing the latest ultra-high performance liquid chromatography-mass spectrometry platform for metabolomics and proteomics research, a diagnostic model for PCOS coexisting with NAFLD was established and evaluated. The 50 patients were randomized 1:1 to receive Canagliflozin/Metformin or Metformin treatment. The Canagliflozin/Metformin group received Canagliflozin 100 mg once daily plus metformin 1000 mg twice daily, and the metformin group received Metformin 1000 mg twice daily, for a continuous period of three months. The study assessed the safety and efficacy of PCOS and NAFLD patients.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-45 years old;
2. Body mass index (BMI) more than 18.5 kg / m2;
3. PCOS diagnosis meets Rotterdam 2003 criteria: at least two of the following symptoms: menstrual menstruation / amenorrhea, hyperandrogenism, and / or biochemical and / or clinical signs of polycystic ovaries.
4. The serum pregnancy test was negative before enrollment.
5. Clinical diagnosis of fatty liver: the ratio of liver to kidney is greater than 1.0.

Can understand the procedures and methods of this clinical trial, patients voluntarily participate and sign the informed consent form, willing to comply with the trial protocol requirements and cooperate with the provision of biological samples for testing as planned.

Exclusion Criteria:

1. Less than 18 years old or more than 45 years old;
2. Patients who are pregnant, intend to become pregnant, are breastfeeding or giving birth;
3. Drug history in the past three months included oral contraceptives, sodium-dependent glucose transporters 2 inhibitors, glucagon-like peptide-1 receptor agonists, thiazolidinediones, metformin, corticosteroids or traditional Chinese medicine.
4. Endocrine disorders such as hyperprolactinemia, thyroid dysfunction and diabetes, Cushing's syndrome, 21-hydroxylase deficiency, congenital adrenal hyperplasia, androgen-secreting tumors, cervical, endometrial or breast cancer.
5. Severe liver function (alanine aminase, aspartate aminase> 3 times normal value or elevation of serum bilirubin to more than 3 times the upper limit of normal) or renal impairment (eGFR <60 ml/min/1.73m2).Severe cardiopulmonary, hematopoietic and hematopoietic insufficiency.
6. Current or past (most recent three months) participation in other studies.
7. Viral hepatitis, autoimmune hepatitis, primary biliary cirrhosis, sclerosing cholangitis, hemochromatosis, anti-trypsin defense, Wilson disease, parenteral nutrition history, use of drugs known to cause steatosis (such as valproate, amiodarone or vitamin E) or liver injury caused by drug abuse.Clinical evidence of hepatic decompensation, such as hepatic encephalopathy, ascites, and variceal bleeding.
8. drank more than 20g per day.
9. Women with persistent or recurrent symptomatic urinary tract infections (UTI), gastrointestinal (GI) problems, or any other condition that may compromise patient safety had strong fertility needs within six months of the study period.
10. Allergic or intolerant to the study drug, unable to continue treatment as required by the protocol, unwilling to complete the study or become pregnant.
11. History of mental illness within 2 years, including any suicidal behavior or major depression, depressive symptoms (defined as Patient Health Questionnaire-9 score more than 15), central nervous system disease (including but not limited to any type of seizure or stroke), and no cognitive behavior (including the investigator considers poor adherence to evaluate efficacy or is unlikely to complete the intended course and follow-up).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-31 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
liver steatosis index CAP (Controlled Attenuation Parameter) measured by FibroScan | at baseline and 12 weeks
  Changes in the liver steatosis index CAP (Controlled Attenuation Parameter) as measured by transient elastography after 12 weeks of treatment.

SECONDARY OUTCOMES:
liver stiffness index (LS） measured by transient elastography, FibroScan | at baseline and 12 weeks
  Changes in the liver stiffness index (LS) (measured by transient elastography) from baseline to 12 weeks of treatment.
Body Composition, including total body water, muscle mass, fat mass (subcutaneous and visceral), fat-free mass detected using Bioelectrical Impedance Analysis (BIA) | at baseline and 12 weeks
  Changes in Body Composition，including total body water, muscle mass, fat mass (subcutaneous and visceral), fat-free mass detected using Bioelectrical Impedance Analysis (BIA) from baseline to 12 weeks of treatment.
selection of proteomics markers using liquid chromatography-tandem mass spectrometry (LC-MS/MS) mass spectrometry for analysis | at baseline and 12 weeks
  Changes in proteomics markers from baseline to 12 weeks of treatment, involving systematic quantification of metabolites and proteins using techniques LC-MS for analysis, with chemometric methods for data interpretation, revealing metabolic pathways and biomarkers.
selection of metabolomics markers by by liquid chromatography-tandem mass spectrometry (LC-MS/MS) mass spectrometryprecision | at baseline and 12 weeks
  Changes in metabolomics markers from baseline to 12 weeks of treatment, including phosphatidylglycerol (PG), Bis(monoacylglycero)phosphate BMP, Sulfatide (sulfatide) (SL), Free fatty acids FFA, Plasmalogen ethanolamine (PE-O), Phosphatidylethanolamine (PE), Phosphatidylinositol (PI), Phosphatidylserine (PS), Monosialosyl ganglioside (GM3) plasmalogen (PCO), Phosphatidylcholine (PC), Lysophosphatidic acid (PA), Lysophosphatidylethanolamine (LPE), Lysophosphatidic acid (LPA), Lysophosphatidylinositol (LPI), Lysophosphatidylserine (LPS), Ceramide(Cer), Lysophosphatidylcholine （LPC), Plasmalogen choline (PCO), Phosphatidylcholine (PC),Sphingomyelin (SM),Sphingosine (Sph）,Ceramide（Cer）,Hexosylceramide （HexCer）, Lactosylceramide （LacCer）, Trihexosylceramide （Gb3), Acylcarnitine acylcarnitine, Monoacylglycerol (MAG), Diglyceride (DAG), Triglyceride (TAG), Cholesteryl ester (CE)
sex hormones by liquid chromatography-tandem mass spectrometry (LC-MS/MS) mass spectrometry | at baseline and after 12 weeks
  Changes in sex hormones by liquid chromatography-tandem mass spectrometry (LC-MS/MS) mass spectrometry from baseline to 12 weeks of treatment, including estriol, hydrocortisone, cortisone, corticosterone, aldosterone, testosterone, 17a-Hydroxyprogesterone, 21-hydroxyprogesterone, DHEA,Estrone, androstenedione, dihydrotestosterone, estradiol,progesterone, pregnenolone, androsterone, epitestosterone, estrone sulfate, estradiol sulfate, epitestosterone sulfate, testosterone sulfate, dhea Sulfate, pregnenolone Monosulfate
Gut Microbiota diversity sequencing by 16s rRNA Amplicon Sequencing Analysis | at baseline and 12 weeks
  Gut microbiome testing equipment includes sterile samplers for sample collection, DNA extraction kits, PCR machines for amplification, high-throughput sequencing platforms for analysis, bioinformatics software for data processing, and AI systems for advanced analysis. These tools enable precise and efficient assessment of gut microbial composition, aiding in understanding its impact on disease and informing clinical treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Li, MD, Study Chair — The First Affiliated Hospital of Shanxi Medical University; Linxin Xu, MD, Principal Investigator — The First Affiliated Hospital of Shanxi Medical University; Yan Wang, Study Director — The First Affiliated Hospital of Shanxi Medical University

REFERENCES:
- [Background] Rocha ALL, Faria LC, Guimaraes TCM, Moreira GV, Candido AL, Couto CA, Reis FM. Non-alcoholic fatty liver disease in women with polycystic ovary syndrome: systematic review and meta-analysis. J Endocrinol Invest. 2017 Dec;40(12):1279-1288. doi: 10.1007/s40618-017-0708-9. Epub 2017 Jun 13. PMID 28612285
- [Background] Makri E, Tziomalos K. Prevalence, etiology and management of non-alcoholic fatty liver disease in patients with polycystic ovary syndrome. Minerva Endocrinol. 2017 Jun;42(2):122-131. doi: 10.23736/S0391-1977.16.02564-5. Epub 2016 Oct 28. PMID 27792214
- [Background] De Sousa SM Dr, Norman RJ Prof. Metabolic syndrome, diet and exercise. Best Pract Res Clin Obstet Gynaecol. 2016 Nov;37:140-151. doi: 10.1016/j.bpobgyn.2016.01.006. Epub 2016 Feb 10. PMID 26972165
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome. Fertil Steril. 2004 Jan;81(1):19-25. doi: 10.1016/j.fertnstert.2003.10.004. PMID 14711538
- [Background] Macut D, Tziomalos K, Bozic-Antic I, Bjekic-Macut J, Katsikis I, Papadakis E, Andric Z, Panidis D. Non-alcoholic fatty liver disease is associated with insulin resistance and lipid accumulation product in women with polycystic ovary syndrome. Hum Reprod. 2016 Jun;31(6):1347-53. doi: 10.1093/humrep/dew076. Epub 2016 Apr 12. PMID 27076501
- [Background] March WA, Moore VM, Willson KJ, Phillips DI, Norman RJ, Davies MJ. The prevalence of polycystic ovary syndrome in a community sample assessed under contrasting diagnostic criteria. Hum Reprod. 2010 Feb;25(2):544-51. doi: 10.1093/humrep/dep399. Epub 2009 Nov 12. PMID 19910321
- [Background] Azziz R, Carmina E, Dewailly D, Diamanti-Kandarakis E, Escobar-Morreale HF, Futterweit W, Janssen OE, Legro RS, Norman RJ, Taylor AE, Witchel SF; Androgen Excess Society. Positions statement: criteria for defining polycystic ovary syndrome as a predominantly hyperandrogenic syndrome: an Androgen Excess Society guideline. J Clin Endocrinol Metab. 2006 Nov;91(11):4237-45. doi: 10.1210/jc.2006-0178. Epub 2006 Aug 29. PMID 16940456
- [Background] Teede HJ, Hutchison SK, Zoungas S. The management of insulin resistance in polycystic ovary syndrome. Trends Endocrinol Metab. 2007 Sep;18(7):273-9. doi: 10.1016/j.tem.2007.08.001. Epub 2007 Aug 16. PMID 17698366
- [Background] Meyer C, McGrath BP, Teede HJ. Overweight women with polycystic ovary syndrome have evidence of subclinical cardiovascular disease. J Clin Endocrinol Metab. 2005 Oct;90(10):5711-6. doi: 10.1210/jc.2005-0011. Epub 2005 Jul 26. PMID 16046590
- [Background] Wild RA, Painter PC, Coulson PB, Carruth KB, Ranney GB. Lipoprotein lipid concentrations and cardiovascular risk in women with polycystic ovary syndrome. J Clin Endocrinol Metab. 1985 Nov;61(5):946-51. doi: 10.1210/jcem-61-5-946. PMID 4044782
- [Background] Mantovani A, Byrne CD, Scorletti E, Mantzoros CS, Targher G. Efficacy and safety of anti-hyperglycaemic drugs in patients with non-alcoholic fatty liver disease with or without diabetes: An updated systematic review of randomized controlled trials. Diabetes Metab. 2020 Nov;46(6):427-441. doi: 10.1016/j.diabet.2019.12.007. Epub 2020 Jan 7. PMID 31923578
- [Background] Itani T, Ishihara T. Efficacy of canagliflozin against nonalcoholic fatty liver disease: a prospective cohort study. Obes Sci Pract. 2018 Aug 22;4(5):477-482. doi: 10.1002/osp4.294. eCollection 2018 Oct. PMID 30338118
- [Background] Cai M, Shao X, Xing F, Zhang Y, Gao X, Zeng Q, Dilimulati D, Qu S, Zhang M. Efficacy of canagliflozin versus metformin in women with polycystic ovary syndrome: A randomized, open-label, noninferiority trial. Diabetes Obes Metab. 2022 Feb;24(2):312-320. doi: 10.1111/dom.14583. Epub 2021 Nov 25. PMID 34726324